CLINICAL TRIAL: NCT06442150
Title: Low-Calorie Medicinal Diet for Type 2 Diabetes Remission: Evaluation of Effectiveness and Exploration of Individual Differences
Brief Title: LCMD for Type 2 Diabetes Remission: Evaluation of Effectiveness and Exploration of Individual Differences
Acronym: LCMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Feng Tao, Director of Endocrinology, Shanghai Municipal Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHMHTCM LCDM
Record Dates: First submitted 2024-05-17; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus in Obese; Type 2 Diabetes
Keywords: Remission of type 2 diabetes; Low Calorie Diet; Medicined Diet; Brain-Gut-Microbiome axis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Due to the unique nature of the intervention, it is not feasible to mask the participants and investigators in the treatment allocation. However, the outcomes assessor will be blinded to minimize potential bias in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCD Group (Active Comparator): Participants will receive a Low-Calorie Diet (815-835 kcal/day; approximately 43% carbohydrate, 29% protein, and 29% fat) meals for 12 weeks, followed by a gradual food reintroduction phase combined with physical activity support for 12 weeks.
  Interventions: Combination Product: Low-Calorie Diet
- LCMD Group (Experimental): Participants will receive a Low-Calorie Medicine Diet (815-835 kcal/day; approximately 43% carbohydrate, 29% protein, and 29% fat) meals product for 12 weeks, followed by a gradual food reintroduction phase combined with physical activity support for 12 weeks.
  Interventions: Combination Product: Low-Calorie Medicine Diet

INTERVENTIONS:
Combination Product: Low-Calorie Medicine Diet — Low-Calorie Medicine Diet meals which are 815-835 kcal/day (approximately 43% carbohydrate, 29% protein, and 29% fat), combined with physical activity.
  Arms: LCMD Group
Combination Product: Low-Calorie Diet — Low-Calorie Diet meals which are 815-835 kcal/day (approximately 43% carbohydrate, 29% protein, and 29% fat), combined with physical activity.
  Arms: LCD Group

SUMMARY:
Type 2 diabetes (T2DM) has become a major public health problem. Achieving remission (HbA1c<6.5% without glucose-lowering medications) has recently become a new treatment goal. Low-calorie diets effectively induce remission, but adverse effects like fatigue, appetite, and constipation hinder success. Integrating traditional Chinese medicine (TCM) herbs into a low-calorie diet may alleviate adverse effects and improve remission rates.

This project investigates the efficacy of a Low-Calorie Medicine Diet (LCMD) in achieving T2DM remission among overweight/obese individuals through a randomized controlled trial. The investigators will explore individual differences in remission and elucidate the underlying biological mechanisms, focusing on the brain-gut-microbiota axis. By integrating nutrition and TCM dietetics, this project provides a novel, evidence-based approach to managing T2DM in Chinese populations.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) has become a major public health problem, and effective prevention and treatment strategies are urgently needed. Recently, the understanding of T2DM has shifted to "a disease that can be remission." Achieving remission, defined as HbA1c<6.5% without using glucose-lowering medications, has become a new treatment goal for T2DM. Evidence suggests that a low-calorie diet is an effective approach to induce remission. Our previous research (NCT05472272) also demonstrated that a low-calorie diet can achieve remission in Chinese T2DM patients.

However, adverse effects during the intervention, such as fatigue, appetite, and constipation, have become significant barriers to successful remission. These symptoms often result in poor adherence to the intervention plan and, consequently, failure to achieve remission. In traditional Chinese medicine (TCM), fatigue and constipation are typical symptoms of "Qi Vacuity", while hunger is more associated with "Yin Vacuity". "Herb is the food" is a unique concept in TCM. Integrating TCM herbs into a low-calorie diet may help alleviate these adverse effects and improve the likelihood of achieving diabetes remission.

This project aims to investigate the efficacy of a Low-Calorie Medicine Diet (LCMD) in achieving remission of T2DM among overweight/obese individuals through a randomized controlled trial. The investigators will also explore individual differences in achieving remission and elucidate the underlying biological mechanisms, focusing on the brain-gut-microbiota axis. By integrating theories from nutrition and TCM dietetics, this project seeks to provide a novel, evidence-based approach to the management of T2DM in Chinese populations.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed T2DM
* The history of T2DM less than 6 years
* Most recent HbA1c higher than 6.5%
* Body mass index: 24-45 kg/m2
* Fasting C-p ≥1.1 ng/ml
* Inability to provide informed consent

Exclusion Criteria:

* Type 1 diabetes, type 2 diabetes currently treated with insulin, or HbA1c ≥12%
* Cardiovascular events within 6 months before trial
* Current use of anti-obesity medications, eating disorders, dieting behaviors, or weight loss >5 kg within 6 months before trial
* Chronic kidney disease stage 3b or above (eGFR <30 mL/min/1.73m²)
* Any condition causing fluid overload, such as heart failure or liver cirrhosis
* Previously diagnosed psychiatric disorders (e.g., schizophrenia, post-traumatic stress disorder, obsessive-compulsive disorder), uncontrolled depression, or epilepsy
* Severe arthritis or active gout
* Active gallstone disease or known as asymptomatic gallstones
* Concurrent enrollment in another clinical trial
* Pregnancy, lactation, or planned conception during the study
* Substance abuse
* Known malignancy
* Comorbidities increasing dietary intervention risk (e.g., biliary disorders)
* Long-term use of antibiotics, corticosteroids, NSAIDs, or PPIs
* Chronic gastrointestinal disorders affecting gut microbiota (e.g., ulcerative colitis)
* Severe hepatic impairment (ALT >2.5× ULN)
* Inability to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving diabetes remission as assessed by American Diabetes Association criteria | Baseline to 24 and 52 weeks
  The proportion of participants achieving diabetes remission, which is defined as having a glycated hemoglobin (HbA1c) level less than 6.5% while receiving no pharmacological therapy for diabetes for at least 3 months.
Number of participants achieving significant weight loss, defined as a reduction of at least 12kg from baseline body weight | Baseline to 12, 24 and 52 weeks
  Proportion of participants achieving significant weight loss (≥12kg/10kg).

SECONDARY OUTCOMES:
Change from baseline in insulin sensitivity as assessed by insulin tolerance test | Baseline to 12, 24 and 52 weeks
  Insulin sensitivity is evaluated with insulin tolerance tests at the pre-specified time points.
Change from baseline in beta cell function as assessed by arginine stimulation test | Baseline to 12, 24 and 52 weeks
  Beta cell function is evaluated with arginine stimulation test at the pre-specified time points.
Change from baseline in liver fat content and pancreatic fat content as assessed by magnetic resonance imaging | Baseline to 12, 24 and 52 weeks
  Liver and pancreatic fat will be assessed using magnetic resonance imaging (MRI) or proton magnetic resonance spectroscopy (1H-MRS). Liver fat content will be quantified as the proton density fat fraction (PDFF) in percentage, while pancreatic fat content will be expressed as the percentage of fat signal relative to the total signal in the region of interest (ROI).
Change from baseline in plasma glucose concentration | Baseline to 12, 24 and 52 weeks
  Glucose homeostasis parameters will be assessed, including fasting blood glucose (FBG) in mmol/L, postprandial blood glucose (PBG) in mmol/L 2 hours after a standardized meal, glycated hemoglobin (HbA1c) in percentage, and time in range (TIR), which represents the percentage of time that blood glucose levels remain within the target range (3.9-10.0 mmol/L) as assessed using continuous glucose monitoring (CGM) or self-monitoring of blood glucose (SMBG).
Change from baseline in fasting serum lipid levels, including total cholesterol, LDL-C, HDL-C, and triglycerides | Baseline to 12, 24 and 52 weeks
  Lipid profile parameters will be assessed, including total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglycerides (TG). All lipid parameters will be measured in mmol/L after at least 8 hours of fasting.
Change from baseline in brain functional connectivity and activity as assessed by functional magnetic resonance imaging | Baseline to 12, 24 and 52 weeks
  Brain functional connectivity and activity will be assessed using functional magnetic resonance imaging (fMRI) during resting state and task-based paradigms. Resting-state fMRI will be used to evaluate the intrinsic functional connectivity among brain regions, focusing on networks related to appetite regulation and cognitive control.
Change from baseline in gut microbiota composition and its metabolites as assessed by 16S rRNA gene sequencing and metabolomics analysis | Baseline to 12, 24 and 52 weeks
  Gut microbiota composition and its metabolites will be assessed through the analysis of fecal samples. 16S rRNA gene sequencing will be used to evaluate gut microbial diversity and composition, focusing on the relative abundance of key bacterial taxa at the phylum, family, and genus levels. Metabolomic profiles, including short-chain fatty acids (SCFAs), bile acids, and amino acids, will be quantified using gas chromatography-mass spectrometry (GC-MS) or liquid chromatography-mass spectrometry (LC-MS).
Change from baseline in the quality of life score as assessed by a validated questionnaire (e.g., SF-36, EQ-5D) | Baseline to 12, 24 and 52 weeks
  Quality of life will be assessed using various validated questionnaires, including the 36-Item Short Form Health Survey (SF-36) for general health status, the EuroQol Five-Dimension (EQ-5D) questionnaire for health-related quality of life, and the Diabetes-Specific Quality of Life (DSQL) questionnaire for diabetes-specific health-related quality of life. The SF-36 and EQ-5D scores range from 0 to 100, with higher scores indicating better health status. The DSQL scores range from 0 to 100, with lower scores indicating better diabetes-specific quality of life.
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 12, 24 and 52 weeks
  Safety will include adverse event incidence, changes in routine blood, urine, and stool tests, alanine transaminase, uric acid, etc. Frequency of constipation and dizziness, as well as scores from PAC-SYM, FSS, FCQ-T, and VAS for hunger, will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Tao, M.D., Principal Investigator — Shanghai Municipal Hospital of Traditional Chinese Medicine
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No